CLINICAL TRIAL: NCT05685134
Title: Invasive and Clinical Features in Patients With Brugada Syndrome Undergoing Catheter Ablation: a Prospective, Single-centre, Randomized, Sham-controlled, and Masked Pilot Study
Brief Title: Invasive and Clinical Features in Patients With Brugada Syndrome Undergoing Catheter Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Mauricio Ibrahim Scanavacca, Director of the Cardiac Arrhythmias Unit; MD, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIS-470
Record Dates: First submitted 2022-12-21; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Brugada Syndrome
Keywords: Brugada syndrome; Radiofrequency catheter ablation; Electroanatomic mapping; Invasive electrophysiological study
MeSH Terms: conditions — Brugada Syndrome | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Prospective, single-centre, randomized, sham-controlled, and masked pilot study with two parallel arms, with a 1:1 allocation ratio to ablation or control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will occur during the electrophysiology procedure, and its automatic computerized process will ensure allocation concealment. The study protocol, for obvious reasons, precludes masking the principal investigator (electrophysiology specialist). Participants randomized to the control group will undergo a sham procedure consisting of femoral venous punctions, catheter insertion, programmed electrical stimulation and electroanatomic mapping, with a similar duration to the ablation procedure. Medical follow-up will be standardized with the same protocol for both treatment groups. All medical documents will be unidentified before being evaluated. Outcome raters and statisticians will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ablation (Experimental): Radiofrequency catheter ablation of the abnormal - prolonged and fragmented - electrophysiologic substrate of Brugada syndrome
  Interventions: Device: Radiofrequency catheter ablation
- Control (Sham Comparator): Femoral venous punctions, catheter insertion, programmed electrical stimulation and electroanatomic mapping, with a similar duration to the ablation procedure
  Interventions: Device: Sham procedure

INTERVENTIONS:
Device: Radiofrequency catheter ablation — Radiofrequency application via catheter to burn the electroanatomic substrate implicated in Brugada syndrome
  Arms: Ablation
Device: Sham procedure — Venous and epicardial punctions, catheter insertions, programmed electrical stimulation and electroanatomical mapping
  Arms: Control

SUMMARY:
This clinical trial aims to learn about the electrophysiological and clinical effects of radiofrequency catheter ablation in patients with Brugada syndrome. The main questions it seeks to answer are:

* What are the immediate effects of catheter radiofrequency ablation in cardiac electrophysiology?
* What is the relation between invasive and clinical features in patients with Brugada syndrome undergoing ablation? Researchers will compare ablation and control groups to see if there is a difference in clinical and invasive markers of the disease in one year of follow-up.

DETAILED DESCRIPTION:
Brugada syndrome (BS) is an electric cardiac disorder characterized by a typical electrocardiographic pattern and an increased risk of cardiac arrhythmias and sudden death. Most arrhythmic events occur during rest, fever or under circumstances of increased vagal activity. In the last decade, catheter ablation has emerged as a valuable and potentially curative therapy for patients with BS. However, little is known about its mechanisms or long-term effects on clinical and invasive markers. This prospective, single-centre, randomized, sham-controlled, and masked pilot study will investigate the impact of catheter ablation in 20 patients with Brugada syndrome, who will be randomized to ablation or control group, with a 1:1 allocation ratio and clinically followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a type 1 Brugada ECG pattern, as characterized by ST-segment elevation (≥2mm) with upward concavity associated with T-wave inversion, in at least one of the right precordial leads, positioned at the second, third or fourth intercostal space, either spontaneously or induced by a provocative test with Class I anti-arrhythmic drugs according to Vaughan Williams
* Patients clinically stable for at least six months before the enrollment
* Able to cope with follow-up visits up to one year after the intervention
* Patients who have signed the written informed consent

Exclusion Criteria:

* Pregnant women
* Patients with structural heart disease
* Patients with a known cardiac or systemic autonomic disorder
* Patients with a history of previous right ventricular outflow tract ablation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Area of abnormal potentials | first 30 minutes after the intervention
  Electroanatomic duration map
Induction of sustained ventricular arrhythmias by programmed electrical stimulation | first 30 minutes after the intervention
  Programmed electrical stimulation (PES) performed on two sites (right ventricular apex and right ventricular outflow tract, unless the patient had inducible ventricular tachycardia at the first location), with energy of twice the diastolic threshold, using two drive cycles (S1: 600 and 430 ms) up to 3 extra stimuli (S2 to S4) with 200 ms as the shortest coupling time. The PVS result is considered positive if sustained ventricular fibrillation or polymorphic ventricular tachycardia is induced.
Maximum potential duration | first 30 minutes after the intervention
  Maximum length of ventricular signs on bipolar electrogram
Local activation time | first 30 minutes after the intervention
  Measured by unipolar catheters placed in the epicardial and endocardial ventricular surfaces
Activation recovery interval | first 30 minutes after the intervention
  Surrogate marker of the action potential duration, measured by unipolar catheters placed in the epicardial and endocardial ventricular surfaces

SECONDARY OUTCOMES:
Spontaneous type 1 Brugada electrocardiographic pattern in standard12 lead and superior leads electrocardiogram | up to one year after the procedure
  Upward ST segment elevation ST-segment elevation ≥2 mm followed by a negative T wave (type 1 Brugada electrocardiographic pattern) in one or more right precordial leads V1 and/or V2 positioned in the second, third, or fourth intercostal spaces.
Spontaneous type 1 Brugada electrocardiographic pattern in 12 lead 24 hour Holter monitoring | up to one year after the procedure
  Upward ST segment elevation ST-segment elevation ≥2 mm followed by a negative T wave (type 1 Brugada electrocardiographic pattern) in one or more right precordial leads V1 and/or V2 positioned in the second, third, or fourth intercostal spaces during 12 lead 24h Holter ECG Monitoring
Spontaneous type 1 Brugada electrocardiographic pattern during treadmill test | up to one year after the procedure
  Upward ST segment elevation ST-segment elevation ≥2 mm followed by a negative T wave (type 1 Brugada electrocardiographic pattern) in one or more right precordial leads V1 and/or V2 positioned in the second, third, or fourth intercostal spaces, during treadmill test.
Occurrence of life threatening arrhythmic events | up to one year after the procedure
  Occurrence of at least one of the following: arrhythmic syncope, documented sustained ventricular tachycardia or ventricular fibrillation, sudden cardiac death or appropriate implantable cardiac defibrillator therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração - InCor - HC/FMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be provided under proper request to the principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the article's publication
Access Criteria: Under request

REFERENCES:
- [Background] Pappone C, Brugada J, Vicedomini G, Ciconte G, Manguso F, Saviano M, Vitale R, Cuko A, Giannelli L, Calovic Z, Conti M, Pozzi P, Natalizia A, Crisa S, Borrelli V, Brugada R, Sarquella-Brugada G, Guazzi M, Frigiola A, Menicanti L, Santinelli V. Electrical Substrate Elimination in 135 Consecutive Patients With Brugada Syndrome. Circ Arrhythm Electrophysiol. 2017 May;10(5):e005053. doi: 10.1161/CIRCEP.117.005053. PMID 28500178
- [Background] Patocskai B, Yoon N, Antzelevitch C. Mechanisms Underlying Epicardial Radiofrequency Ablation to Suppress Arrhythmogenesis in Experimental Models of Brugada Syndrome. JACC Clin Electrophysiol. 2017 Apr;3(4):353-363. doi: 10.1016/j.jacep.2016.10.011. Epub 2016 Dec 21. PMID 28948234
- [Background] Kotake Y, Barua S, Kazi S, Virk S, Bhaskaran A, Campbell T, Bennett RG, Kumar S. Efficacy and safety of catheter ablation for Brugada syndrome: an updated systematic review. Clin Res Cardiol. 2023 Dec;112(12):1715-1726. doi: 10.1007/s00392-022-02020-3. Epub 2022 Apr 22. PMID 35451610